CLINICAL TRIAL: NCT06264232
Title: A Multi-center, Prospective, Randomized, Controlled Clinical Trial to Demonstrate the Safety and Effectiveness of the Full Visual Range AT ELANA 841P Posterior Chamber Intraocular Lens for Correction of Aphakia Following Cataract Removal
Brief Title: AT ELANA 841P Posterior Chamber Intraocular Lens for Correction of Aphakia Following Cataract Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT ELANA 841P-BER-303-24
Record Dates: First submitted 2024-02-12; First posted 2024-02-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-02

CONDITIONS: Cataract Senile
Keywords: Cataract; Cataract Surgery
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking will include not knowing which type of IOLs were received by the subject until end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- AT ELANA 841P IOL (Experimental): Cataract Surgery to implant multifocal intraocular lenses
  Interventions: Device: Cataract Surgery
- CT LUCIA 621P IOL (Active Comparator): Cataract Surgery to implant monofocal intraocular lenses
  Interventions: Device: Cataract Surgery

INTERVENTIONS:
Device: Cataract Surgery — Bilateral removal of age related cataractous lenses with the implantation of intraocular lenses to improve visual acuity.

SUMMARY:
The goal of this clinical trial is to demonstrate the safety and effectiveness of the full visual range AT ELANA 841P IOL when used to treat adult patients having cataract surgery. Subjects will be randomly selected to receive a pair of IOLs, either the AT ELANA 841P or CT LUCIA 621P lens design. All patients will undergo surgery in both eyes, and they will receive follow up care for up to 6-months. During this time, all patients will undergo thorough eye exams at every study visit and complete questionnaires about their quality of vision post-surgery.

DETAILED DESCRIPTION:
The goal of this clinical trial is to demonstrate safety and effectiveness of the full visual range AT ELANA 841P posterior chamber IOL when used to treat adult patients undergoing cataract surgery. In this study, all patients will be randomly assigned (using a 1 to 1 ratio) to receive either the investigational device: AT ELANA 841P trifocal IOL, or the commercially available, FDA-approved, control device: CT LUCIA 621P monofocal IOL.

There will be 286 adults, 22 years of age or older. All will be scheduled to undergo cataract surgery in both eyes; along with completing a 6-months follow-up. This clinical trial will take place at 14 clinical sites located throughout the United States.

Salus IRB will provide ethical oversight for this clinical trial, while Ora, Inc. is the CRO assisting the research sites with completing all required study activities.

This clinical trial is expected to be about 18-months long.

Each participant who provides their consent for study participation must meet the following visual criteria to qualify:

* Before Cataract Surgery: Best-Corrected Visual Acuity 20/40 or worse with or without glare present.
* Astigmatism of 1.0 diopter or less in both eyes
* After Cataract Surgery: Best-Corrected Visual Acuity is expected to be better than 20/30

Study Enrollment is anticipated to begin June 2024, and will last about 10-months. During this time, subjects will undergo cataract surgery in both eyes, and after surgery will attend about 8 follow-up visits spread over 6-months. At these visits each individual will have their vision thoroughly examined, and be asked to complete questionnaires about the quality of their vision.

Typical Assessments each participant will have at their study visits include:

* You will be asked about your current overall health and about any previous conditions or treatments you have had.
* Any medications you have taken, are taking now or have stopped taking while in the study will be recorded.
* Visual acuity and Subjective refraction (glasses prescription): your doctor will test your far vision with and without glasses.
* Biometry: the anatomy of your eye will be measured using a specialized instrument to calculate the recommended IOL power for your eyes.
* Pupil diameter: the study doctor will measure the size of your pupils.
* Intraocular pressure: numbing drops will be put in your eyes and your eye pressure will be measured by touching an instrument to your cornea, which is the clear front window of your eye. Since your eyes are numb, you should feel no pain during this procedure.
* Slit lamp examination: the front part of your study eye will be examined using a bright light and a special microscope called a slit lamp. Dilating drops could be put in your study eye to enlarge your pupil (the black circle in the center of the colored part [the iris] of the eye). The study doctor will use a magnifying lens and a bright light to examine your retina, which is the back of your eye. The effect of these drops will last approximately 4 -5 hours, and during that time, it is recommended that you should not drive a car or operate machinery.
* Dilated fundus (retina) examination: once the pupil is dilated, the study doctor will observe the back part of your eyes.
* Questionnaire: you will be asked to complete a questionnaire to collect information on any problems which involve your vision or feelings that you have about the condition of your vision.

Later in the study, these assessments will be performed for each participant:

* Contrast Sensitivity: a special device will be used to test how well you can differentiate objects on a bright background with different lighting conditions (Month 6 only).
* Defocus Curve: your study doctor will place different lenses in front of your eyes. This simulates how you would see at different distances without changing your position to the test chart. Your vision will be measured to determine how well you are able to see at each of the distances (Month 1, Month 6).

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 22 years of age or older at the time of study enrollment
2. Bilateral cataractous lens changes as demonstrated by best corrected distance visual acuity of 0.30 logMAR (20/40) or worse either with or without a glare source present (e.g., Brightness Acuity Tester) for which phacoemulsification cataract extraction and posterior chamber IOL implantation is indicated
3. Best corrected distance visual acuity projected to be better than 0.20 logMAR (better than 20/30) after cataract removal and IOL implantation
4. Preoperative keratometric (corneal) astigmatism of 1.00 D or less (≤1.00 D) in both operative eyes
5. Clear intraocular media other than cataract
6. Contact lens wear is to be discontinued two (2) weeks for soft contact lenses both daily and extended wear; and ≥ 30 days for rigid gas permeable lenses prior to preoperative biometry and keratometry testing.
7. Calculated lens power within the available range
8. Subject is willing to sign the IRB-approved informed consent form
9. Subject is willing, able and has sufficient cognitive awareness to comply with examination procedures and schedule for follow-up visits

Exclusion Criteria:

1. Presence of systemic disease that could increase the operative risk or confound the outcome, including but not limited to diabetes mellitus, active cancer treatment, mental illness, dementia, immunocompromised, connective tissue disease, clinically significant atopic disease, etc.
2. Ocular condition that may predispose for future complications, including but not limited to dry eye syndromes or symptoms, anterior segment pathology, glaucoma (uncontrolled despite intake of medication), history of cystoid macular edema, macular degeneration as confirmed by clinical examination and adjunct testing (e.g., OCT, FA)
3. Clinically significant corneal abnormalities, including corneal dystrophy (epithelial, stromal or endothelial dystrophy), irregularity, inflammation or edema; conditions including but not limited to active/inactive keratitis, keratoconjunctivitis, kerato uveitis, keratopathy, keratectasia
4. Previous intraocular or corneal surgery that might confound the outcome of the investigation or increase the risk to the subject, including corneal transplants, retinal detachment, glaucoma surgeries, refractive laser procedures including but not limited to LASIK, limbal relaxing incision, Small Incision Lenticule Extraction (SMILE) etc.
5. Use of or history of use of systemic medications with significant ocular side effects or any medications that could confound the outcome or increase subject risk (e.g., Tamsulosin Hydrochloride [Flomax] or other medications including anticholinergics or alpha-adrenergic blocking agents with similar side effects [e.g., small pupil/floppy iris syndrome], antimetabolites, etc.)
6. Currently taking systemic steroids and/or planned on taking systemic steroids prior to operative visit and during the course of the investigation.
7. Subjects with diagnosed degenerative visual disorders, including but not limited to macular degeneration or other retinal disorders (such as diabetic retinopathy, diabetic macular edema, retinal detachment) that are predicted to confound outcomes or to cause future acuity loss to 0.20 logMAR or worse.
8. Subjects with conditions that increase the risk of zonular rupture (e.g., pseudoexfoliation syndrome, Marfan's syndrome) during cataract extraction procedure that may affect the postoperative centration or tilt of the IOL
9. Expected concomitant ocular procedure during cataract surgery or within the next 12 months (e.g., glaucoma surgery including implantation of MIGS, astigmatic correction surgery, penetrating keratoplasty [PK], laser-assisted in situ keratomileusis, SMILE etc.)
10. Subjects who are expected to require retinal laser treatment within the next 12 months
11. History of amblyopia or monofixation syndrome with poor stereoscopic vision
12. Rubella, congenital, traumatic or complicated cataracts
13. History of or current anterior or posterior segment inflammation, including but not limited to iritis or uveitis
14. Microphthalmos or macrophthalmos
15. Iris defects (e.g., aniridia)
16. Optic nerve atrophy
17. Keratoconus or Irregular astigmatism, as determined by topography
18. Inability to perform keratometry, topography or biometry (including but not limited to cataract density, subject unable to focus for longer time etc.) or subjects with unstable keratometry, topography or biometry measurements
19. Pathologic miosis caused by anterior segment pathology in the study eye (e.g., chronic uveitis, iritis, rubeosis iridis, neurological conditions such as multiple sclerosis, Argyle Robertson's pupil, acquired or congenital Horner´s syndrome, etc.)
20. Pupil diameter less than 6 mm when fully dilated
21. Pregnant, lactating at time of enrollment, or has another condition with associated fluctuation of hormones that could lead to refractive changes
22. Subject whose freedom is impaired by administrative or legal order
23. Concurrent participation in another drug or device investigation that could confound the outcome of this investigation
24. Subjects unable to achieve keratometry stability after discontinuing contact lens wear
25. Gonioscopic abnormalities

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Outcome | Month 6
  Mean, monocular photopic logMAR best-corrected distance visual acuity (BCDVA) at 4 m for the first implanted eyes, at Month 6 (Visit 4).
Primary Effectiveness Outcome | Month 6
  Mean, monocular photopic logMAR distance-corrected near visual acuity (DCNVA) at 40 cm, for the first implanted eyes at Month 6 (Visit 4)
Primary Effectiveness Outcome | Month 6
  Mean, monocular photopic logMAR distance-corrected intermediate visual acuity (DCIVA) for the first implanted eyes at 66 cm, at Month 6 (Visit 4)
Primary Effectiveness Outcome | Month 6
  Mean, monocular photopic logMAR distance-corrected visual acuity (DCVA) at 1 m (equal to -1 D defocus) and 50 cm (equal to -2 D defocus), for the first implanted eyes at Month 6 (Visit 4)
Primary Effectiveness Outcome | Month 6
  Proportion of AT ELANA 841P IOL eyes achieving monocular photopic BCDVA 0.30 logMAR or better, for first implanted eyes in Full Analysis Set (FAS) and Best Case Set (BCS), at Month 6 (Visit 4)
Primary Safety Outcome | Month 6
  Mean log monocular mesopic far contrast sensitivity (without glare at spatial frequency of 1,5, 3, 6, and 12 cycles/degree) for first implanted eyes in Best Case Set (BCS), at Month 6 (Visit 4)
Primary Safety Outcome | Month 6
  Rate of secondary surgical interventions related to the optical properties of the lens for first implanted eyes, through 6 months.
Primary Safety Outcome | Month 6
  Rate of Posterior Chamber IOL cumulative and persistent adverse events (AEs) listed in the ISO 11979-7:2024 Table E.2, for first implanted eyes, through 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Seth M Pantanelli, MD, Principal Investigator — Penn State Health
Locations (14):
- United States (14):
  - Beverly Hills Institute of Ophthalmology, Beverly Hills, California
  - Mitchell C Shultz MD/Shultz Chang Vision, Northridge, California
  - Coastal Vision Medical Group, Orange, California
  - Cape Coral Eye Center, Cape Coral, Florida
  - Chu Vision Institute, Bloomington, Minnesota
  - Ophthalmology Consultants of St Louis, St Louis, Missouri
  - Vance Thompson Vision-Nebraska, Omaha, Nebraska
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina
  - Vance Thompson Vision-South Dakota, Sioux Falls, South Dakota
  - Whitsett Vision Group, Houston, Texas
  - Texas Eye & Laser, Hurst, Texas
  - PNV Clinical Research, San Antonio, Texas
  - Eye Centers of Racine & Kenosha, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No